CLINICAL TRIAL: NCT05876247
Title: Speech Flexibility in Adulthood Following Oral Cancer Treatment: Acoustic and Kinematic Explorations
Brief Title: Articulatory Adaptation Following Oral Cancer Treatment
Acronym: SPOKE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: METc 2021/711
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Speech Disorders
Keywords: Articulation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Speech Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals treated for oral cancer: Dutch native speakers (18+) who will undergo surgical treatment for a T1 or T2 tumour on the tongue.
  Interventions: Other: Electromagnetic Articulography
- Control speakers: Dutch native speakers (18+) without self-reported speech problems.
  Interventions: Other: Electromagnetic Articulography

INTERVENTIONS:
Other: Electromagnetic Articulography — Motion tracking sensors will track articulatory movements of the tongue, jaw and lips

SUMMARY:
The goal of this longitudinal study is to learn more about the articulatory consequences of surgical oral cancer treatment. The main aims are to study the coordination and development of speech articulation of patients who will undergo surgical treatment for oral cancer longitudinally and whether individual differences in the reliance on auditory or tactile information can predict the success of speech compensatory strategies.

Participants will perform multiple speech tasks while motion tracking sensors track the articulatory gestures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with T1 or T2 tumor in the oral cavity
2. At least 18 years old and able to provide informed consent
3. Native speaker of Dutch
4. Has nog been treated for oral cancer before

Exclusion Criteria:

1a. Recurrence of disease (for patients)

1b. Treated for oral cancer (for healthy controls) 2. Speech problems (e.g., stuttering) 3. Problems with sight or hearing that impede reading or understanding instructions. When glasses or a hearing aid resolve these problems, then participants are not excluded.

4. Neurological or psychological disorders (e.g., stroke) 5. Non-removable metal in, on or around the head (piercings, braces, pacemaker, electrodes) 6. Self-reported signs of depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with and without oral cancer who speak Dutch as their native language
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Articulatory gestures | 2022-2025
  Articulatory movements in three dimensions of the tongue, lips and jaw as measured by the NDI Vox Electromagnetic Articulograph. Measures include: articulator speed (mm/s), total displacement (mm), coordinates (x,y,z) during specific gestures.
Acoustic outcomes | 2022-2025
  Speech acoustics will be measured in Praat and include the first and second formants of vowels (in Hz), global movement size in terms of acoustic working space (Hz-squared), and the centre of gravity of sibilants (in Hz)

CONTACTS AND LOCATIONS:
Overall Officials: Max Witjes, PhD, Principal Investigator — University of Groningen
Locations (2):
- Netherlands (2):
  - Faculty of Arts, University of Groningen, Groningen
  - University Medical Centre Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Will share where legally possible.